CLINICAL TRIAL: NCT00352807
Title: Absorption of Brimonidine Ophthalmic Solution in the Aqueous Humor of Cataract Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Allergan (Industry)
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0501-45
Record Dates: First submitted 2006-07-14; First posted 2006-07-17 (Estimated); Last update posted 2007-10-17 (Estimated); Status verified 2007-10

CONDITIONS: Cataract
Keywords: Cataract
MeSH Terms: conditions — Cataract | interventions — Brimonidine Tartrate

INTERVENTIONS:
Drug: Brimonidine Purite

SUMMARY:
The purpose of this study is to obtain and assay human aqueous samples following pre-operative dosing with 0.1% Brimonidine Purite™ (pH 7.8) or with 0.15% Brimonidine Purite® (pH 7.2) from patients undergoing routine cataract surgery in order to evaluate the aqueous concentration of the two formulations.Study hypothesis: The aqueous humor concentration 45 minutes following dosing of 0.1% Brimonidine Purite™ (pH 7.8) is comparable with 0.15% Brimonidine Purite® (pH 7.2)

DETAILED DESCRIPTION:
The purpose of this study is to obtain and assay human aqueous samples following pre-operative dosing with 0.1% Brimonidine Purite™ (pH 7.8) or with 0.15% Brimonidine Purite® (pH 7.2) from patients undergoing routine cataract surgery in order to evaluate the aqueous concentration of the two formulations.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must:

  1. Be willing and able to provide written Informed Consent
  2. Be able and willing to follow instructions and likely to complete the entire course of the study.
  3. Be male or female of any race at least 18 years of age.
  4. Have visually significant cataract for which they have elected to undergo cataract surgery.

Exclusion Criteria:

* No subject may:

  1. Known allergy or sensitivity to the study medication or its components
  2. Contraindications to brimonidine therapy: concurrent use of monoamine oxidase (MAO) inhibitor therapy
  3. Have any active ocular disease other than glaucoma or ocular hypertension that would interfere with study parameters (such as: uveitis, ocular infection, or severe dry eye). Patients with mild chronic blepharitis, age-related macular degeneration, background diabetic retinopathy may be enrolled at the discretion of the investigator.
  4. Any ocular surgery (including laser, refractive, intraocular filtering surgery, or any other ocular surgery) within 3 months.
  5. Require use of ocular medications (including glaucoma medications), except intermittent use of artificial tears.
  6. Have corneal abnormalities that would interfere with the ability to obtain an adequate sample safely or have a shallow anterior chamber which would make obtaining an aqueous sample difficult at the time of surgery in the opinion of the investigator.
  7. Be concurrently enrolled in an investigational drug or device study or participation within the last 30 days in any investigational drug or device study.
  8. Be pregnant, nursing, planning a pregnancy, or be of childbearing potential and not using a reliable form of contraception.
  9. Have a situation or condition that in the investigator's opinion may put the subject at significant risk, may confound the study results, or may interfere significantly with participation in the study such as, significant cardiovascular disease, hepatic or renal impairment, depression, Raynaud's, orthostatic hypotension; uncontrolled high blood pressure. or concomitant use of other potential CNS depressants and tricyclics, (Amendment 1, May 25, 2005)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22
Dates: Start 2005-02; Study Completion 2005-12

PRIMARY OUTCOMES:
Bioanalysis of brimonidine concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Louis B Cantor, MD, Principal Investigator — IUPUI/Clarian
Locations (4):
- United States (4):
  - University Hospital, Indianapolis, Indiana
  - Veterans Affairs Medical Center, Indianapolis, Indiana
  - Wishard Memorial Hospital, Indianapolis, Indiana
  - Iu Eye at Carmel, Indianapolis, Indiana

REFERENCES:
- [Background] PK-02-P027 Relative ocular bioavailability of 0.2% Alphagan and 0.15% Brimonidine-BAK to that of 0.15% Alphagan P in female albino rabbits. Allergan 2002.
- [Background] PK-02-P041 Comparison of ocular and systemic bioavailability of three 0.10% brimonidine purite formulations to that of 0.15% Alphagan P in albino rabbits. Allergan 2002.